CLINICAL TRIAL: NCT01147991
Title: A Phase I, Dose Escalation Trial of Recombinant Modified Vaccinia Ankara (MVA)-Based Vaccine Encoding Epstein-Barr Virus Target Antigens
Brief Title: Vaccine Therapy in Treating Patients With Epstein-Barr Virus-Related Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000675266; CRUK-PH1-101; EUDRACT-2004-001931-46
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Gastric Cancer; Head and Neck Cancer; Lymphoma; Lymphoproliferative Disorder; Nonneoplastic Condition
Keywords: Epstein-Barr virus infection; stage I nasopharyngeal cancer; stage II nasopharyngeal cancer; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; post-transplant lymphoproliferative disorder; stage I gastric cancer; stage II gastric cancer; adult nasal type extranodal NK/T-cell lymphoma; angioimmunoblastic T-cell lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Stomach Neoplasms; Head and Neck Neoplasms; Lymphoma; Lymphoproliferative Disorders; Epstein-Barr Virus Infections; Nasopharyngeal Neoplasms; Hodgkin Disease; Lymphoma, Extranodal NK-T-Cell; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic

INTERVENTIONS:
Biological: EBNA1 C-terminal/LMP2 chimeric protein-expressing recombinant modified vaccinia Ankara vaccine
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with Epstein-Barr virus and cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine safety and to characterize the toxicity profile of EBNA1 C-terminal/LMP2 chimeric protein-expressing recombinant modified vaccinia Ankara vaccine in patients in remission having been treated conventionally for Epstein-Barr virus (EBV) and malignancy.
* To describe changes in the frequency of functional T-cell responses to major histocompatibility complex (MHC) class I and II-restricted epitopes within EBNA1 and LMP2 in peripheral blood at sequential time-points before, during, and up to nine months after the vaccination course in these patients.

Secondary

* To assess changes in levels of EBV genome in plasma in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive EBNA1 C-terminal/LMP2 chimeric protein-expressing recombinant modified vaccinia Ankara vaccine intradermally on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for immune function, biomarker, and pharmacological studies.

After completion of study treatment, patients are followed up at weeks 11 and 14, and at 6 months and 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy of a type typically associated with Epstein-Barr virus (EBV) latent infection meeting the following criteria:

  * The presence of EBV within the malignant cells has been demonstrated by immunohistochemistry for viral antigens or by EBER (EBV early RNA) in situ hybridization
* Patients in remission from disease or with disease for which no standard treatment is appropriate, as defined by 1 of the following groups:

  * Have achieved a continuing complete response (CR) or unconfirmed CR
  * Residual masses at the site of treated disease that are not progressing (i.e., stable disease) and for which no standard therapy is recognized
  * Residual or recurrent disease that is low-volume and causing minimal or no symptoms and for which no standard therapy is recognized
* Completed standard therapy for malignancy ≥ 12 weeks before trial entry

  * No more than 1 course of chemotherapy as treatment for EBV+ malignancy
* No ongoing toxic manifestations of prior treatment, except alopecia or certain grade 1 toxicities at the discretion of the investigator and Cancer Research UK
* No patients with active EBV+ cancer for whom evidence-based active treatment is available and likely to be offered to prolong life or relieve symptoms within 14 weeks of the first vaccination

PATIENT CHARACTERISTICS:

* WHO performance status 0 or 1
* Life expectancy ≥ 4 months
* Lymphocyte count must satisfy 1 of the following criteria:

  * Greater than lower limit of the reference range in the investigator site
  * Greater than or equal to 0.5 x 10^9/L AND recovery from nadir of lymphocyte numbers following primary treatment for EBV+ malignancy, judged by no successive rises in lymphocyte count measured up to 3 successive occasions 3 weeks apart
* Hemoglobin > 10.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum alkaline phosphatase < 1.5 times ULN
* ALT and/or AST < 1.5 times ULN
* Calculated creatinine clearance > 50 mL/min (uncorrected value) OR isotope clearance measurement > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for 6 months after completion of study treatment
* No known chronic active infection with hepatitis B, hepatitis C, or HIV
* No history of anaphylaxis or severe allergy to vaccinations
* No allergy to eggs or egg products
* No ongoing active infection
* No known splenic dysfunction
* No concurrent active autoimmune disease
* No prior NYHA class III or IV cardiac disease or concurrent congestive heart failure
* No concurrent active skin diseases requiring therapy (i.e., psoriasis, eczema)
* No other condition that, in the Investigator's opinion, would make the patient not a good candidate for this clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior myeloablative therapy followed by an autologous or allogeneic hematopoietic stem cell transplant
* More than 12 weeks since prior and no concurrent chemotherapy or radiotherapy
* No splenectomy or splenic irradiation
* No concurrent immunosuppressive medication, including corticosteroids

  * Long-term prophylactic use of inhaled corticosteroids allowed
* No major thoracic and/or abdominal surgery within the past 4 weeks from which the patient has not yet recovered
* No other concurrent anticancer or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of drug-related grade 3 or 4 systemic or local adverse events (defined using the NCI CTCAE version 3.0)
Occurrence of local skin reactions considered related to the vaccination
Occurrence of drug-related systemic reactions (e.g., transient fever)
Demonstration by ELIspot assays of the frequency of T-lymphocytes recognizing major histocompatibility complex (MHC) class I and II-restricted epitopes within EBNA1 and LMP2 in peripheral blood at sequential time-points before, during, and up to 9 mo ...

SECONDARY OUTCOMES:
Measurement of EBV-genome levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Neil M Stevens, MD, Principal Investigator — University of Birmingham
Locations (3):
- United Kingdom (3):
  - University of Birmingham, Birmingham, England
  - Royal Marsden - London, London, England
  - Christie Hospital, Manchester, England